CLINICAL TRIAL: NCT04290104
Title: Is an Antibiotic Prescription Required After Laparoscopic Cholecystectomy for Acute Calculous Cholecystitis?
Brief Title: Is an Antibiotic Prescription Required After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, principal investigator, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSU Konya HPRC
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Cholecystitis; Acute, With Cholelithiasis
Keywords: cholecystectomy; antibiotic
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Intervention Model Description: Patients discharged after laparoscopic cholecystectomy for acute Calculous Cholecystitis constitutes the study population. The patients discharged are randomized into two groups by the clinical secretary with the help of a computer program.
  Antibiotics are included in the prescription given to group 1 on the way home. The patient receives 1 gram of Ampicillin/sulbactam twice daily for 5-7 days at home.
  The patient, who was randomized to the second group, does not have antibiotics on his prescription.
  After the patients are discharged, they are called for weekly control for a month, and they are examined in terms of surgical site infection.
  The study reaches the result by making statistical analysis in terms of the rate of surgical site infection between both groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1gr oral ampicillin/sulbactam group (Experimental): The group to be prescribed 1 g oral ampicillin/sulbactam twice a day while discharged after laparoscopic cholecystectomy due to ACC.
  Interventions: Drug: 1gr oral ampicillin/sulbactam group
- Antibiotic not prescribed group (No Intervention): Antibiotics not prescribed when discharged after laparoscopic cholecystectomy due to ACC.

INTERVENTIONS:
Drug: 1gr oral ampicillin/sulbactam group — Group prescribed 1 g oral ampicillin/sulbactam 2 times a day.
  Arms: 1gr oral ampicillin/sulbactam group

SUMMARY:
The need for antibiotics to reduce surgical site infection after cholecystectomy for acute calculous cholecystitis is still controversial. The researchers aimed to investigate the effect of antibiotics prescribed on surgical site infection when discharged to patients undergoing laparoscopic cholecystectomy for acute calculous cholecystitis.

DETAILED DESCRIPTION:
Cholecystectomy is the definitive treatment for acute calculous cholecystitis (ACC). In the past, the timing of cholecystectomy has been the subject of debate. Early cholecystectomy performed within 72 hours at the beginning of the disease is preferred to first medical treatment and delayed cholecystectomy 6 to 10 weeks after recovery. In many studies, it suggests early cholecystectomy because it provides a definitive solution, faster recovery times, and more rapid return to work.

Surgical site infections (SSIs) are a significant cause of mortality and morbidity after surgery. In the United States alone, more than 300,000 surgical field infections are seen annually. Again, in the United States alone, the budget spent on surgical site infection reaches $ 10 billion. Antibiotic treatment in ACC patients to prevent surgical site infection is a standard practice in the hospital before and after surgery. However, there is controversy over the use of antibiotics to prevent surgical site infection after discharge. The researchers aimed to investigate the effect of antibiotics prescribed on surgical site infection when discharged to patients undergoing laparoscopic cholecystectomy (LC) for acute calculous cholecystitis.

Patients and Method Patients who were admitted to the General Surgery Clinic with the diagnosis of acute calculous cholecystitis and who underwent early Laparoscopic Cholecystectomy will be included in the study. Patients will be told in detail about the study protocol, and those who accept it will be included in the study. A study consent form, which is written and signed by patients in their handwriting, will be taken. The patients will be staged as Stage 1,2,3 according to the TG13 criteria accepted at the Tokyo 2013 consensus. The anesthesiologist will make ASA classification. Oral intake of the patients will be stopped, and parenteral fluid and anti biotherapy will be applied. The demographic characteristics, comorbidities of the patients, will be recorded in their files, whether they had previous ACC attacks. Patients will be operated within 12-72 hours after hospitalization. Amoxycillin / sulbactam 1 g will be administered parenterally three times a day to patients before and after surgery. Patients included in the post-operative study will be discharged within three days at the latest if the complication has not developed. Just before discharge, the clinical secretary will give a code to each patient with the help of a computer program, and block randomization will be made and divided into two groups. Those who received oral antibiotics (AB group) and those who did not receive antibiotics (HA group).

The primary purpose of antibiotic therapy in ACC is to limit both systemic septic response and local inflammation to prevent SSI in the superficial wound, fascia, and organ cavity. In this study, ampicillin/sulbactam will be used according to the TG18 guidelines (according to recommendation). If the patient is in the AB group, 1 g of ampicillin/sulbactam will be prescribed two times a day and will use for a total of 5-7 days. All demographic features and medical processes of the patients will be recorded electronically with the hospital medical computer program (Deva Data ®).

If SSI is detected by clinical examination and other diagnostic methods (laboratory, ultrasound, and tomography), the antibiotic regimen will be changed in the AB group, and ampicillin/sulbactam will be started in the NA group. Also, superficial and deep SSI will locally be drained, organ SSI will be drained by ultrasonography or tomography-guided.

Sample size calculation: As the reported rate of postoperative SSIs associated with ACC varies between 1% and 15%, it was estimated that 102 patients per group would allow detecting a 10% difference in the rate of complications with 80% power with a confidence interval of 5%. The estimated price of loss to follow-up was 10%; therefore, at least 112 patients were needed to be enrolled for each group.

ELIGIBILITY:
Inclusion Criteria:

* Acute calculous cholecystitis patients over the age of 18 will be included.

Exclusion Criteria:

* Laparoscopic cholecystectomy patients who have been elective for symptomatic cholelithiasis,
* Patients who are hospitalized with ACC and who undergo late LC, have decompensated systemic disease,
* Patients with ASA 4,
* Patients who underwent surgery for early LC due to ACC diagnosis and left laparoscopic method for reasons such as difficult dissection and underwent open cholecystectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
surgical site infections | one month
  The development of SSI in the operational area or other parts of the body is considered the primary outcome. All patients will be followed up for a postoperative month. It is classified as incisional SSI, CDC guidelines, and superficial, deep, and organ infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Magill SS, Edwards JR, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Survey of health care-associated infections. N Engl J Med. 2014 Jun 26;370(26):2542-3. doi: 10.1056/NEJMc1405194. No abstract available. PMID 24963580
- [Background] Duncan CB, Riall TS. Evidence-based current surgical practice: calculous gallbladder disease. J Gastrointest Surg. 2012 Nov;16(11):2011-25. doi: 10.1007/s11605-012-2024-1. Epub 2012 Sep 18. PMID 22986769